CLINICAL TRIAL: NCT02927067
Title: A Phase 3, Multicenter, Randomized, Double-blind, Double-dummy, Active-controlled Study to Assess the Efficacy and Safety of Maribavir Compared to Valganciclovir for the Treatment of Cytomegalovirus (CMV) Infection in Hematopoietic Stem Cell Transplant Recipients
Brief Title: A Study of Maribavir Compared to Valganciclovir to Treat Cytomegalovirus Infections in People Who Have Received Stem Cell Transplants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP620-302; 2015-004726-34 (EudraCT Number)
Record Dates: First submitted 2016-09-29; First posted 2016-10-06 (Estimated); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Cytomegalovirus (CMV)
MeSH Terms: interventions — maribavir; Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Valganciclovir 900 mg BID (Active Comparator): Participants received 900 milligrams (mg) of valganciclovir along with a placebo matched to maribavir, twice daily (BID) orally for 8 weeks. Valganciclovir dose was allowed to be adjusted to 450 mg BID or 450 mg QD based on renal function impairment assessed at baseline or development of neutropenia during the study.
  Interventions: Drug: Valganciclovir; Other: Placebo
- Maribavir 400 mg BID (Experimental): Participants received 400 mg of maribavir along with a placebo matched to valganciclovir, BID orally for 8 weeks.
  Interventions: Drug: Maribavir; Other: Placebo

INTERVENTIONS:
Drug: Maribavir — Participants will receive 400 mg of maribavir BID orally.
  Arms: Maribavir 400 mg BID
Drug: Valganciclovir — Participants will receive valganciclovir tablets orally.
  Arms: Valganciclovir 900 mg BID
Other: Placebo — Participants will receive placebo tablets matched to either maribavir or valganciclovir.

SUMMARY:
This study is about treatment options for cytomegalovirus infections in people who have received stem cell transplants. The main aim of the study is to check if the cytomegalovirus infection can no longer be detected after treatment with marivabir or valganciclovir.

Participants will take 2 tablets of marivabir or valganciclovir and 2 tablets of placebo twice a day for 8 weeks. A placebo will look like marivabir or valganciclovir but will not have any medicine in it.

After treatment, each participant will be followed up for up to 12 weeks.

Participants will visit their study clinic up to 18 times during the study.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide written, personally signed, and dated informed consent to participate in the study before completing any study-related procedures. As applicable, a parent/both parents or legally authorized representative (LAR) must provide signature of informed consent and there must be documentation of assent by the participants before completing any study-related procedures. During the COVID-19 public health emergency, informed consent from a potential or current trial participant may, if permitted by local laws and regulations, be obtained via electronic informed consent (eIC) capabilities or an electronic face-to-face consent interview when these individuals are unable to travel to the site (FDA COVID-19 Guidance, 27 January 2021, Q11).
* Be greater than or equal to (>=) 16 years of age at the time of consent.
* Be a recipient of hematopoietic stem cell transplant.
* Have a documented asymptomatic CMV infection, with a screening value of CMV DNA >=1365 International Units per millilitre (IU/mL) to less than or equal to (<=) 273000 IU/mL in whole blood or >=455 IU/mL to <=91000 IU/mL in plasma in 2 consecutive assessments, separated by at least 1 day, as determined by local or central specialty laboratory quantitative polymerase chain reaction (qPCR) or comparable quantitative CMV DNA results. Both samples should be taken within 14 days prior to randomization with second sample obtained within 5 days prior to randomization. Same laboratory and same sample type (whole blood or plasma) should be used for these assessments. Asymptomatic CMV infection is defined as an infection that does not present with tissue invasive CMV disease, as assessed by the investigator. Participants with CMV DNA less than (<) 910 and >=455 IU/mL in plasma or <2730 and >=1365 IU/mL in whole blood will also need to meet at least 1 of the following criteria for high-risk CMV infection to be eligible:

  1. Human leukocyte antigen (HLA)-related (sibling) donor with at least 1 mismatch at 1 of the following 3 HLA-gene loci: HLA-A, -B or -DR,
  2. Haploidentical donor
  3. Unrelated donor with at least 1 mismatch at 1 of the following 4 HLA -gene loci: HLA-A, -B, -C and -DRB1,
  4. Use of umbilical cord blood as stem cell source,
  5. Use of ex vivo T-cell-depleted grafts,
  6. Grade 2 or greater graft-versus-host-disease (GVHD), requiring the use of systemic corticosteroids (defined as the use of >=1 milligram per kilogram per day (mg/kg/day) of prednisone or equivalent dose of another corticosteroid).
* Have the current CMV infection as the first episode of CMV viremia after HSCT, either primary or reactivation, which in the investigator's opinion requires treatment.
* Per investigator's judgment, be eligible for treatment with valganciclovir.
* Have all of the following results as part of screening laboratory assessments (results from either the central laboratory or a local laboratory can be used for qualification):

  1. Absolute neutrophil count to >=1000 per cubic millimeter (/mm^3) [1.0*10^9/L].
  2. Platelet count >=25,000/mm^3 [25*10^9/L].
  3. Hemoglobin >=8 grams per deciliter (g/dL).
  4. Estimated creatinine clearance >=30 milliliters per minute (mL/min).
* Have a negative serum beta human chorionic gonadotropin (beta-HCG) pregnancy test at screening, if a female of child bearing potential. Urine pregnancy tests may be done per institutional requirements; however they are not sufficient for eligibility determination. Sexually active females of child bearing potential must agree to comply with any applicable contraceptive requirements of the protocol. If male, must agree to use an acceptable method of birth control, as defined in the protocol, during the study treatment administration period and for 90 days afterward the last dose of study treatment.
* Be able to swallow tablets.
* Have life expectancy of >=8 weeks.
* Weigh >=40 kilograms (kg).
* Be willing and have an understanding and ability to fully comply with study procedures and restrictions defined in the protocol.

Exclusion Criteria:

* Have CMV tissue invasive disease as assessed by the investigator at the time of screening and randomization at Visit 2/Day 0.
* Have a CMV infection that is known to be genotypically resistant to ganciclovir, valganciclovir, foscarnet, or cidofovir based on documented evidence.
* Be presenting with recurrent CMV infection (defined as a new detection of CMV infection in a participants who had at least one previously documented episode of CMV infection post-transplant, and who has had at least 2 weeks of undetectable CMV DNA between the episodes during active surveillance, based on same local laboratory and same sample type). The Participants must also have been off any anti-CMV treatment between the current and prior infection. Otherwise, the current infection may be considered continuation of the prior infection.
* Require ganciclovir, valganciclovir, foscarnet, or cidofovir administration for conditions other than CMV when study treatment is initiated (example: herpes simplex virus [HSV] co-infection requiring use of any of these agents after the randomization) or would need a co-administration with maribavir for CMV infection.
* Be receiving leflunomide, letermovir, or artesunate when study treatment is initiated.

Note: Participants who may be receiving leflunomide must discontinue the use at least 14 days prior to randomization at Visit 2/Day 0 and the first dose of study treatment. Participants receiving letermovir must discontinue use 3 days prior to first dose of study treatment. Participants receiving artesunate must discontinue the use prior to the first dose of study treatment.

* Be on treatment with anti-CMV agents (ganciclovir, valganciclovir, foscarnet or letermovir) for the current CMV infection for longer than 72 hours.
* Have known hypersensitivity to the active substance or to an excipient of the study treatments.
* Have severe vomiting, diarrhea, or other severe gastrointestinal illness within 24 hours prior to the first dose of study treatment that would preclude administration of oral medication.
* Require mechanical ventilation or vasopressors for hemodynamic support at the time of randomization.
* Be female and pregnant or nursing.
* Have previously completed, discontinued, or have been withdrawn from this study.
* Have received any investigational agent with known anti-CMV activity within 30 days before initiation of study treatment or CMV vaccine at any time.
* Have received any unapproved agent or device within 30 days before initiation of study treatment.
* Have any clinically significant medical or surgical condition that, in the investigator's opinion, could interfere with interpretation of study results, contraindicate the administration of the assigned study treatment, or compromise the safety or well-being of the participant.
* Have previously received maribavir.
* Have serum aspartate aminotransferase (AST) greater than (>) 5 times upper limit of normal (ULN) at screening, or serum alanine aminotransferase (ALT) >5 times ULN at screening, or total bilirubin >= 3.0*ULN at screening (except for documented Gilbert's syndrome), as analyzed by local or central laboratory.
* Have known (previously documented) positive results for human immunodeficiency virus (HIV). Participants must have a confirmed negative HIV test result within 3 months of study entry or, if unavailable, be tested by a local laboratory during the screening period.
* Have active malignancy with the exception of nonmelanoma skin cancer, as determined by the investigator. Participants who experience relapse or progression of their underlying malignancy (for which HSCT was performed), as determined by the investigator, are not to be enrolled.
* Be undergoing treatment for acute or chronic hepatitis C

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (129):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - Colorado Blood Cancer Institute - PPDS, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - PIN, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Joan and sandford I. Weill Medical College of Cornell University Clinic, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Saint Davids South Austin Medical Center, Austin, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - VA Puget Sound Health Care System - NAVREF - PPDS, Seattle, Washington
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - Medizinische Universitat Wien (Medical University of Vienna), Vienna, Vienna
  - Elisabethinen Hospital Linz, Linz
- Belgium (8):
  - UZ Antwerpen, Edegem, Antwerpen
  - Institute Jules Bordet, Brussels, Brussels Capital
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - Universitair Ziekenhuis Brussel - PIN, Jette, Brussels Capital
  - University Hospital Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
  - AZ Sint-Jan AV, Bruges, West-Vlaanderen
  - CHU de Liège, Liège
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
- China (8):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Xiangya Hospital Central South University, Changsha
  - Guangzhou First People's Hospital, Guangzhou
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- University Hospital Center Zagreb, Zagreb, Croatia
- Czechia (2):
  - Fakultni nemocnice v Motole, Prague, Praha, Hlavní Mesto
  - Ustav hematologie a krevni transfuze, Prague
- France (13):
  - Institut de Cancérologie Strasbourg Europe, Strasbourg, Bas-Rhin
  - Hopital de Hautepierre, Strasbourg, Bas-Rhin
  - CHU de Bordeaux, Pessac, Gironde
  - Hôpital Universitaire Dupuytren, Limoges, Haute-Vienne
  - CHU de GRENOBLE, Grenoble, Isère
  - Hôtel Dieu, Nantes, Loire-Atlantique
  - CHU Angers, Angers, Maine-et-Loire
  - Hopital Henri Mondor, Créteil, Val-de-Marne
  - Hopital Jean Minjoz, Besnçon
  - Institut Paoli Calmettes, Nice
  - Hôpital Saint Antoine, Paris
  - Hôpital Saint Louis, Paris
  - EDOG - Institut Claudius Regaud - PPDS, Toulouse
- Germany (11):
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universität des Saarlandes, Homburg, Saarland
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Universitätsklinikum Augsburg, Augsburg
  - Helios Klinikum Berlin-Buch, Berlin
  - Martin Luther Universitat Halle Wittenberg, Halle
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Universitätsklinik Rostock, Rostock
  - Robert Bosch Krankenhaus, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
- Greece (2):
  - Attikon University General Hospital, Athens, Attica
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Del-pesti Centrumkorhaz- Orszagos Hematologiai és Infektologiai Intezet, Budapest, Hungary
- Israel (4):
  - Sheba Medical Center - PPDS, Ramat Gan, Central District
  - Hadassah Medical Center - PPDS, Jerusalem, Jerusalem
  - Rambam Medical Center - PPDS, Haifa
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Italy (7):
  - Ospedale Dell'Angelo, Brescia, Lombardy
  - Ospedale Infantile Regina Margherita - INCIPIT - PIN, Turin, Piedmont
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona, Veneto
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione Policlinico Universitario A Gemelli, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- New Zealand (2):
  - Auckland City Hospital, Grafton, Auckland
  - Canterbury Health Laboratories, Christchurch, South Island
- Poland (3):
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - MTZ Clinical Research Sp z o o - PRATIA - PPDS, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
- Russia (3):
  - First St. Petersburg State Medical University n.a. I.P Pavlov, Saint Petersburg, Sankt-Peterburg
  - Regional Oncology Center, Irkutsk
  - Kirov Research Institute of Haematology and Blood Transfusion, Kirov
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital (SGH), Singapore
- South Korea (2):
  - Dong-A University Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
- Spain (14):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca, Castille and León
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - ICO l'Hospitalet Hospital Duran i Reynals, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga
  - Hospital Universitario de Donostia, San Sebastian Gipuzkoa
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Universitätsspital Zürich, Zurich, Switzerland
- Turkey (Türkiye) (2):
  - Baskent University Medical Faculty Adana Practice and Research Center, Adana
  - Ankara University Medica Faculty Hematology Department Clinical Research Area PPDS, Ankara
- United Kingdom (7):
  - Birmingham Heartlands Hospital, West Midlands, Birmingham
  - Hammersmith Hospital, London, London, City of
  - University College London, London, London, City of
  - St George's Hospital, Tooting, London
  - Clatterbridge Cancer Centre Liverpool, Liverpool, Merseyside
  - The Christie NHS Foundation Trust - PPDS, Manchester
  - Southampton University Hospitals NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Chou S, Winston DJ, Avery RK, Cordonnier C, Duarte RF, Haider S, Maertens J, Peggs KS, Solano C, Young JH, Gu J, Pocock G, Papanicolaou GA. Comparative Emergence of Maribavir and Ganciclovir Resistance in a Randomized Phase 3 Clinical Trial for Treatment of Cytomegalovirus Infection. J Infect Dis. 2025 Mar 17;231(3):e470-e477. doi: 10.1093/infdis/jiae469. PMID 39302855
- [Derived] Papanicolaou GA, Avery RK, Cordonnier C, Duarte RF, Haider S, Maertens J, Peggs KS, Solano C, Young JH, Fournier M, Murray RA, Wu J, Winston DJ; AURORA Trial Investigators. Treatment for First Cytomegalovirus Infection Post-Hematopoietic Cell Transplant in the AURORA Trial: A Multicenter, Double-Blind, Randomized, Phase 3 Trial Comparing Maribavir With Valganciclovir. Clin Infect Dis. 2024 Mar 20;78(3):562-572. doi: 10.1093/cid/ciad709. PMID 38036487
- [Derived] Stewart AG, Kotton CN. What's New: Updates on Cytomegalovirus in Solid Organ Transplantation. Transplantation. 2024 Apr 1;108(4):884-897. doi: 10.1097/TP.0000000000004855. Epub 2023 Oct 30. PMID 37899366
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd74db2bf003ab46ecf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 97 sites in United States,Spain,France,Germany,United Kingdom,Belgium,China,Italy,Israel,Australia,Canada,Singapore,Croatia, Czech Republic,Greece,Hungary,Korea,New Zealand,Poland,Russia,Switzerland, and Turkey from 14 April 2017(first participant first visit) to 01 July 2022(last participant last visit).
Pre-assignment Details: Participants who were hematopoietic stem cell transplant (HSCT) recipients with a diagnosis of asymptomatic cytomegalovirus (CMV) infection were enrolled then randomized in a 1:1 ratio to receive either maribavir or valganciclovir (along with placebo matched to comparator) in each arm in a double-blind, double-dummy fashion.
Period: Overall Study
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Started | 277 | 276
Treated Participants (Treated participants (full analysis set) included the participants from the randomized set who took at least one dose of assigned study drug and were analyzed for efficacy and safety evaluations.) | 274 | 273
Participants Received 8 Weeks Treatment (Participants who received 8 weeks of treatment include the participants who completed study drug treatment.) | 140 | 179
Completed | 217 | 215
Not Completed | 60 | 61
Not completed — Withdrawn Consent | 20 | 12
Not completed — Death | 18 | 31
Not completed — Adverse Event | 13 | 10
Not completed — Noncompliance | 5 | 2
Not completed — Reason not Specified | 4 | 6

BASELINE CHARACTERISTICS:
Population: Randomized set included all participants in the enrolled set for whom a randomization number had been assigned.
Groups:
- Valganciclovir 900 mg BID: Participants received 900 mg of valganciclovir along with a placebo matched to maribavir, BID orally for 8 weeks. Valganciclovir dose was allowed to be adjusted to 450 mg BID or 450 mg QD based on renal function impairment assessed at baseline or development of neutropenia during the study.
- Total: Total of all reporting groups
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID | Total
Number analyzed (Participants) | 277 | 276 | 553
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (15.22) | 53.1 (13.96) | 52.5 (14.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 126 | 236
  Male | 167 | 150 | 317
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 35 | 72
  Not Hispanic or Latino | 193 | 216 | 409
  Unknown or Not Reported | 47 | 25 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 39 | 36 | 75
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 9 | 10 | 19
  White | 200 | 221 | 421
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 9 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 13 | 19 | 32
  China | 9 | 9 | 18
  Korea, South | 3 | 2 | 5
  New Zealand | 10 | 7 | 17
  Belgium | 31 | 30 | 61
  Switzerland | 4 | 2 | 6
  Czech Republic | 0 | 2 | 2
  Germany | 9 | 11 | 20
  Spain | 61 | 69 | 130
  France | 34 | 14 | 48
  United Kingdom | 14 | 14 | 28
  Greece | 1 | 0 | 1
  Croatia | 4 | 4 | 8
  Hungary | 2 | 1 | 3
  Israel | 2 | 2 | 4
  Italy | 7 | 4 | 11
  Poland | 1 | 2 | 3
  Russia | 1 | 0 | 1
  Turkey | 6 | 5 | 11
  Canada | 8 | 7 | 15
  United States | 50 | 61 | 111
  Singapore | 7 | 11 | 18
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is the number of participants with data available for analysis for height.
  cm
    number analyzed (Participants) | 264 | 267 | 531
    (all) | 169.58 (9.391) | 168.75 (9.579) | 169.17 (9.486)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed is the number of participants with data available for analysis for weight.
  kg
    number analyzed (Participants) | 270 | 275 | 545
    (all) | 70.31 (15.247) | 70.98 (16.779) | 70.65 (16.027)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI = Body Mass Index. It is computed by [weight (kg) / height (cm)^2] x 10,000. Population: Number analyzed is the number of participants with data available for analysis for BMI.
  kg/m^2
    number analyzed (Participants) | 263 | 266 | 529
    (all) | 24.38 (4.628) | 24.90 (5.007) | 24.64 (4.825)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Confirmed Clearance of Plasma Cytomegalovirus (CMV) Deoxyribose Nucleic Acid (DNA) at the End of Study Week 8
Description: Confirmed CMV viremia clearance is defined as plasma CMV DNA concentrations less than lower limit of quantification (LLOQ; i.e. <137 International units per milliliter [IU/mL]), when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV Test in 2 consecutive post baseline samples separated by at least 5 days. To be considered a responder for the primary endpoint, the participant must have received exclusively study-assigned treatment (regardless of whether study-assigned treatment was completed).
Time Frame: Week 8
Population: Modified randomized set (i.e., the full analysis set) included all participants in the randomized set who took at least 1 dose of assigned study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Number analyzed (Participants) | 274 | 273
Participants | 212 | 190
Statistical Analysis 1: Comparison: Valganciclovir 900 mg BID vs Maribavir 400 mg BID; Test type: Non-Inferiority — Non-inferiority (NI) margin of primary efficacy endpoint was 7%. If lower limit of 95% confidence interval (CI) was greater than -7%, NI was assumed. Power calculation: Assuming 68% (maribavir), 60% (valganciclovir) participants achieve confirmed viremia clearance,494 participants (247 per group) would yield >90% power to declare NI based on 2-group test of equivalence in proportions. Considering 10% dropout,550 participants (275 per group) were planned to be enrolled and randomized; Difference in Percentage of Responders = -7.7, 95% CI 2-sided [-14.98 to -0.36] — Cochran-Mantel-Haenszel (CMH) weighted average approach (stratified for baseline plasma CMV DNA concentration and acute GVHD status) was used for adjusted difference in percentage of responders (Maribavir-Valganciclovir), 95% CI, and p-value

2. Secondary Outcome: Number of Participants Who Achieved Confirmed CMV Viremia Clearance and CMV Infection Symptom Control at the End of Week 8, Followed by Maintenance of Treatment Effect at Week 16
Description: Confirmed CMV viremia clearance is defined as plasma CMV DNA concentrations less than lower limit of quantification (LLOQ; i.e. <137 International units per milliliter [IU/mL]), when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV Test in 2 consecutive post baseline samples separated by at least 5 days. To be considered a responder for this key secondary endpoint, the participant must have received exclusively study-assigned treatment (regardless of whether study-assigned treatment was completed). CMV Infection Symptom Control is defined as no new clinical findings of CMV tissue invasive disease. Maintenance of Treatment Effect is defined as maintaining confirmed CMV viremia clearance and CMV infection symptom control through Week 16.
Time Frame: Week 8 up to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Number analyzed (Participants) | 274 | 273
Participants | 133 | 144
Statistical Analysis 1: Comparison: Valganciclovir 900 mg BID vs Maribavir 400 mg BID; Test type: Non-Inferiority — The non-inferiority margin of the key secondary efficacy endpoint was 7%. If the lower limit of the 95% CI was greater than -7%, then noninferiority (NI) was assumed. Because the NI of the primary efficacy endpoint was not established, the NI hypothesis of the key secondary endpoint was not tested formally; Difference in Percentage of Responders = 4.4, 95% CI 2-sided [-3.91 to 12.76] — CMH weighted average approach (stratified for baseline plasma CMV DNA concentration and acute GVHD status) was used for the adjusted difference in percentage of responders (Maribavir-Valganciclovir), the corresponding 95% CI, and the p-value

3. Secondary Outcome: Number of Participants Who Achieved Confirmed Clearance of Plasma CMV DNA (CMV Viremia Clearance) at Week 8 After Receiving 8 Weeks of Study Assigned Treatment
Description: Confirmed CMV viremia clearance is defined as plasma CMV DNA concentrations less than lower limit of quantification (LLOQ; i.e. <137 International units per milliliter [IU/mL]), when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV Test in 2 consecutive post baseline samples separated by at least 5 days. To be considered a responder for this secondary endpoint, the participant must have received exclusively study-assigned treatment for 8 weeks. Participants who discontinued treatment early were non-responders for this endpoint.
Time Frame: Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Number analyzed (Participants) | 274 | 273
Participants | 137 | 158
Statistical Analysis 1: Comparison: Valganciclovir 900 mg BID vs Maribavir 400 mg BID; Test type: Superiority; p = 0.061, Cochran-Mantel-Haenszel — The CMH weighted average approach (stratified for baseline plasma CMV DNA concentration and acute GVHD status) was used for the adjusted difference in percentage of responders (Maribavir-Valganciclovir), the corresponding 95% CI, and the p-value; Difference in Percentage of Responders = 8.0, 95% CI 2-sided [-0.38 to 16.30]

4. Secondary Outcome: Number of Participants Who Achieved Confirmed CMV Viremia Clearance After Receiving 8 Weeks of Study-assigned Treatment Through Weeks 12, 16 and 20
Description: Confirmed CMV viremia clearance is defined as plasma CMV DNA concentrations less than lower limit of quantification (LLOQ; i.e. <137 International units per milliliter [IU/mL]), when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV Test in 2 consecutive post baseline samples separated by at least 5 days. To be considered a responder for this secondary endpoint, the participant must have received exclusively study-assigned treatment for 8 weeks.
Time Frame: Week 8 through Weeks 12, 16 and 20
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Number analyzed (Participants) | 274 | 273
Participants
  Week 8 | 137 | 158
  Week 12 | 98 | 134
  Week 16 | 82 | 119
  Week 20 | 72 | 98
Statistical Analysis 1: Comparison: Valganciclovir 900 mg BID vs Maribavir 400 mg BID; Week 8; Test type: Superiority; p = 0.061, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference in Percentage of Responders = 8.0, 95% CI 2-sided [-0.38 to 16.30]
Statistical Analysis 2: Comparison: Valganciclovir 900 mg BID vs Maribavir 400 mg BID; Week 12; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference in Percentage of Responders = 13.4, 95% CI 2-sided [5.23 to 21.62]
Statistical Analysis 3: Comparison: Valganciclovir 900 mg BID vs Maribavir 400 mg BID; Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference in Percentage of Responders = 13.8, 95% CI 2-sided [5.80 to 21.87]
Statistical Analysis 4: Comparison: Valganciclovir 900 mg BID vs Maribavir 400 mg BID; Week 20; Test type: Superiority; p = 0.014, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference in Percentage of Responders = 9.7, 95% CI 2-sided [1.98 to 17.50]

5. Secondary Outcome: Number of Participants Who Maintained Confirmed CMV Viremia Clearance at Week 8 After Receiving Study-Assigned Treatment Through Study Weeks 12 and 20 Regardless of Whether Study Assigned Treatment Was Completed
Description: Confirmed CMV viremia clearance is defined as plasma CMV DNA concentrations less than lower limit of quantification (LLOQ; i.e. <137 International units per milliliter [IU/mL]), when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV Test in 2 consecutive post baseline samples separated by at least 5 days. To be considered a responder for this secondary endpoint, the participant must have received exclusively study-assigned treatment (regardless of whether the 8-week study-assigned treatment was completed or discontinued early) and had no symptoms of tissue invasive CMV disease at Week 8, Week 8 through Week 12, and Week 8 through Week 20, respectively.
Time Frame: Week 8 through Weeks 12 and 20
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Number analyzed (Participants) | 274 | 273
Participants
  Week 8 | 211 | 190
  Week 12 | 157 | 162
  Week 20 | 116 | 118
Statistical Analysis 1: Comparison: Valganciclovir 900 mg BID vs Maribavir 400 mg BID; Week 8; Test type: Superiority; p = 0.051, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference in Percentage of Responders = -7.3, 95% CI 2-sided [-14.64 to 0.02]
Statistical Analysis 2: Comparison: Valganciclovir 900 mg BID vs Maribavir 400 mg BID; Week 12; Test type: Superiority; p = 0.606, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference in Percentage of Responders = 2.2, 95% CI 2-sided [-6.05 to 10.37]
Statistical Analysis 3: Comparison: Valganciclovir 900 mg BID vs Maribavir 400 mg BID; Week 20; Test type: Superiority; p = 0.809, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference in Percentage of Responders = 1.0, 95% CI 2-sided [-7.27 to 9.31]

6. Secondary Outcome: Number of Participants With Confirmed Recurrence of Viremia During First 8 Weeks of the Study
Description: Recurrence of CMV viremia is defined as plasma CMV DNA concentration greater than or equal to (>=) lower limit of quantification (LLOQ, i.e. >=137 International units per milliliter [IU/mL]) when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV Test in 2 consecutive plasma samples at least 5 days apart, after being unquantifiable (<LLOQ, i.e. <137 IU/mL) for at least 5 days in 2 consecutive samples during the first 8 weeks of the study, during the 12 weeks of the follow up study phase, and at any time during the study.
Time Frame: Up to Week 8
Population: Overall number analyzed is the subset of participants from the modified randomized set (all participants in the randomized set who took at least 1 dose of study-assigned treatment) who achieved confirmed viremia clearance.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Number analyzed (Participants) | 236 | 226
Participants | 6 | 16

7. Secondary Outcome: Number of Participants With Confirmed Recurrence of Viremia During the Follow-up Period
Description: Recurrence of CMV viremia is defined as plasma CMV DNA concentration greater than or equal to (>=) LLOQ when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV Test in 2 consecutive plasma samples at least 5 days apart, after being unquantifiable (<LLOQ) for at least 5 days in 2 consecutive samples during the first 8 weeks of the study, during the 12 weeks of the follow up study phase, and at any time during the study.
Time Frame: From Week 9 up to Week 20
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Number analyzed (Participants) | 236 | 226
Participants | 47 | 27

8. Secondary Outcome: Number of Participants With Confirmed Recurrence of Viremia at Any Time During the Study
Description: as for outcome 7
Time Frame: Up to Week 20
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Number analyzed (Participants) | 236 | 226
Participants | 53 | 43

9. Secondary Outcome: Number of Participants With Confirmed Recurrence of Viremia While on Study Treatment and Off Treatment
Description: as for outcome 7
Time Frame: Baseline up to Week 20
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Number analyzed (Participants) | 236 | 226
Participants
  On Study Treatment | 0 | 14
  Off Study Treatment | 53 | 29

10. Secondary Outcome: Number of Participants With Grade 3 or 4 (Shift From Baseline Grade <3) and Grade 4 Neutropenia (Shift From Baseline Grade <4) While on Study Treatment
Description: Grade 3 and grade 4 neutropenia are defined as absolute neutrophil count (ANC) <1000 per cubic millimeter (/mm^3) and ANC <500/mm^3 respectively. Incidence of Grade 3 or 4 neutropenia represents the percentage of participants with Grade <3 (or missing) neutropenia at baseline, but Grade 3 or 4 while on study treatment. Incidence of Grade 4 neutropenia represents the number of participants with Grade <4 (or missing) neutropenia at baseline, but Grade 4 while on study treatment.
Time Frame: From start of study drug to end of study drug + 1 day (up to approximately Week 8)
Population: Safety set included all participants who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Number analyzed (Participants) | 274 | 273
Participants
  Grade 3 or Grade 4 Neutropenia | 137 [44.08 to 55.92] | 44 [11.76 to 20.48]
  Grade 4 Neutropenia | 61 [17.34 to 27.19] | 9 [1.18 to 5.41]

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events During the On-Treatment Period
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participants administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE that has a start date on or after the first dose of study treatment, or that has a start date before the date of first dose of study treatment but increases in severity after the first dose of study treatment, will be considered a treatment-emergent AE (TEAE).
Time Frame: From the start of the study treatment to 7 days after the last dose of study treatment (up to approximately Week 9)
Population: Safety set included all participants who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Number analyzed (Participants) | 274 | 273
Participants | 269 | 268

12. Secondary Outcome: Predose Concentration (Cmin) of Maribavir
Description: The primary plasma maribavir concentration dataset (primary concentration dataset) includes all plasma maribavir concentrations. Missing PK sampling times are imputed according to the sparse sampling schedule in primary concentration dataset.
Time Frame: Weeks 1, 4, and 8: pre-morning dose
Population: Pharmacokinetic (PK) Set included all participants in the safety set who received maribavir treatment and had plasma samples drawn and tested for maribavir concentrations. Overall number analyzed is the number of participants available for analyses. Number analyzed is the number of participants available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Maribavir 400 mg BID
Number analyzed (Participants) | 225
micrograms per milliliter (µg/mL)
  Week 1 | 9.17 (7.69)
  Week 4: number analyzed (Participants) | 190
  Week 4 | 8.71 (9.20)
  Week 8: number analyzed (Participants) | 164
  Week 8 | 7.02 (6.35)

13. Secondary Outcome: Area Under the Concentration-Time Curve Over the 12-Hour Dosing Interval at Steady State AUC(0-tau) of Maribavir for Adolescent Participants Only
Time Frame: Pre-morning dose, 1, 2, 3, 4, 6, 8, and 12 hours post-morning dose of Week 1
Population: An adolescent PK set consisted of all participants of ≥16 to <18 years of age in the safety set who received maribavir treatment and had plasma samples drawn and tested for maribavir concentrations. Overall number analyzed is the number of participants available for analyses.
Measure: Mean (Full Range); unit: hours (h)*μg/mL
Arm/Group | Maribavir 400 mg BID
Number analyzed (Participants) | 1
hours (h)*μg/mL | 161 [161 to 161]

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Maribavir for Adolescent Participants Only
Time Frame: Pre-morning dose, 1, 2, 3, 4, 6, 8, and 12 hours post-morning dose of Week 1
Population: as for outcome 13
Measure: Mean (Full Range); unit: µg/mL
Arm/Group | Maribavir 400 mg BID
Number analyzed (Participants) | 1
µg/mL | 22.0 [22.0 to 22.0]

15. Secondary Outcome: Time When Maximum Concentration is Observed (Tmax) of Maribavir for Adolescent Participants Only
Time Frame: Pre-morning dose, 1, 2, 3, 4, 6, 8, and 12 hours post-morning dose of Week 1
Population: as for outcome 13
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Maribavir 400 mg BID
Number analyzed (Participants) | 1
hours (h) | 0.92 [0.92 to 0.92]

16. Secondary Outcome: Apparent Oral Clearance (CL/F) of Maribavir for Adolescent Participants Only
Time Frame: Pre-morning dose, 1, 2, 3, 4, 6, 8, and 12 hours post-morning dose of Week 1
Population: as for outcome 13
Measure: Mean (Full Range); unit: liters per hour (L/h)
Groups:
- Maribavir 400 mg BID: Participants received 400 mg of maribavir along with a placebo matched to valganciclovir; BID orally for 8 weeks.
Arm/Group | Maribavir 400 mg BID
Number analyzed (Participants) | 1
liters per hour (L/h) | 2.49 [2.49 to 2.49]

17. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Maribavir for Adolescent Participants Only
Time Frame: Pre-morning dose, 1, 2, 3, 4, 6, 8, and 12 hours post-morning dose of Week 1
Population: as for outcome 13
Measure: Mean (Full Range); unit: liters (L)
Arm/Group | Maribavir 400 mg BID
Number analyzed (Participants) | 1
liters (L) | 18.3 [18.3 to 18.3]

18. Other Pre Specified Outcome: Number of Participants Developing Resistance
Description: Resistance was defined as the presence of any CMV resistance-associated amino acid substitution that has been documented (or suspected) to be associated with reduced susceptibility to conventional anti-CMV therapies (ganciclovir/valganciclovir, foscarnet, and cidofovir) or maribavir. Genotypic resistance analyses were restricted to sequence variants that were known or suspected to be associated with resistance to conventional anti-CMV therapies or maribavir as of January 21, 2022. A participant was categorized as having developed resistance if the central lab genotyping results indicated the presence of one or more treatment-emergent resistance mutations.
Time Frame: From start of study drug up to end of the study (up to Week 20)
Population: Safety set included all participants who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
Number analyzed (Participants) | 274 | 273
Participants | 8 | 24

ADVERSE EVENTS:
Time Frame: All-cause mortality: From start of study drug up to end of the study (up to Week 20); Serious and Other Adverse Events: From the start of the study drug to 7 days after the last dose of study treatment (up to approximately Week 9)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Valganciclovir 900 mg BID | Maribavir 400 mg BID
All-Cause Mortality (participants affected / at risk) | 29/277 | 37/276
Serious Adverse Events (participants affected / at risk) | 95/274 | 88/273
Other Adverse Events (participants affected / at risk) | 256/274 | 245/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valganciclovir 900 mg BID (N=274) | Maribavir 400 mg BID (N=273)
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Acute graft versus host disease in intestine (Immune system disorders) | 4 | 10
Acute graft versus host disease in skin (Immune system disorders) | 1 | 4
Acute graft versus host disease oral (Immune system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Acute polyneuropathy (Nervous system disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Chronic graft versus host disease (Immune system disorders) | 1 | 0
Chronic graft versus host disease in eye (Immune system disorders) | 0 | 1
Chronic graft versus host disease in intestine (Immune system disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 5 | 2
Cystitis viral (Infections and infestations) | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 2
Cytomegalovirus enterocolitis (Infections and infestations) | 1 | 0
Cytomegalovirus gastritis (Infections and infestations) | 1 | 0
Cytomegalovirus gastroenteritis (Infections and infestations) | 1 | 0
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 3 | 3
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 2
Cytomegalovirus oesophagitis (Infections and infestations) | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 4 | 1
Device related infection (Infections and infestations) | 1 | 1
Device related sepsis (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Disseminated toxoplasmosis (Infections and infestations) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Dysbiosis (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dysuria (Renal and urinary disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 2
Epstein-Barr viraemia (Infections and infestations) | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 2
Eye infection toxoplasmal (Infections and infestations) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 1
Fournier's gangrene (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Fungal sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis astroviral (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Herpes zoster disseminated (Infections and infestations) | 0 | 1
Herpes zoster meningoencephalitis (Infections and infestations) | 0 | 2
Herpes zoster reactivation (Infections and infestations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 2
Infection (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Leukaemic infiltration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Limbic encephalitis (Nervous system disorders) | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Neurosensory hypoacusis (Ear and labyrinth disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Nystagmus (Nervous system disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 2
Parainfluenzae virus infection (Infections and infestations) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 3
Pneumonia cytomegaloviral (Infections and infestations) | 2 | 1
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Product use issue (Injury, poisoning and procedural complications) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 13 | 8
Renal impairment (Renal and urinary disorders) | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 3
Shock (Vascular disorders) | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Syncope (Nervous system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 4
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Toxoplasmosis (Infections and infestations) | 0 | 1
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transplant rejection (Immune system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1
Warm type haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valganciclovir 900 mg BID (N=274) | Maribavir 400 mg BID (N=273)
Abdominal pain (Gastrointestinal disorders) | 19 | 14
Acute graft versus host disease in skin (Immune system disorders) | 32 | 46
Anaemia (Blood and lymphatic system disorders) | 49 | 62
Asthenia (General disorders) | 19 | 13
Blood creatinine increased (Investigations) | 12 | 18
Constipation (Gastrointestinal disorders) | 10 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 20
Decreased appetite (Metabolism and nutrition disorders) | 16 | 18
Diarrhoea (Gastrointestinal disorders) | 44 | 50
Dysgeusia (Nervous system disorders) | 16 | 47
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 2
Fatigue (General disorders) | 19 | 13
Headache (Nervous system disorders) | 14 | 30
Hypertension (Vascular disorders) | 17 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 22 | 23
Leukopenia (Blood and lymphatic system disorders) | 27 | 7
Nausea (Gastrointestinal disorders) | 64 | 74
Neutropenia (Blood and lymphatic system disorders) | 144 | 44
Neutrophil count decreased (Investigations) | 29 | 13
Oedema peripheral (General disorders) | 26 | 27
Platelet count decreased (Investigations) | 16 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 10
Pyrexia (General disorders) | 25 | 24
Renal impairment (Renal and urinary disorders) | 15 | 24
Taste disorder (Nervous system disorders) | 6 | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 62 | 31
Tremor (Nervous system disorders) | 15 | 10
Vomiting (Gastrointestinal disorders) | 47 | 55
White blood cell count decreased (Investigations) | 14 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT02927067/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT02927067/SAP_001.pdf